CLINICAL TRIAL: NCT01361880
Title: Randomized Messaging Trial to Reduce African-American Infant Mortality
Brief Title: Reduce African-American Infant Mortality
Acronym: SIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Children's National Research Institute (Other); Medstar Health Research Institute (Other)
Responsible Party: Principal Investigator, Rachel Moon, MD, Principal Investigator, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2011-095
Record Dates: First submitted 2011-05-12; First posted 2011-05-27 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-06

CONDITIONS: Health Behavior
Keywords: African American; Anticipatory Guidance; Health Promotion; Infant Mortality; Injury Prevention; Nurses; Parent Education; sudden Infant Death Syndrome
MeSH Terms: conditions — Health Behavior; Infant Death; Sudden Infant Death | interventions — Health Promotion; Infant Mortality; Nurses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Reduce infant mortality (Other): The overall purpose of this study is to develop and evaluate a systematic approach to improve African-American parental behaviors specifically with regards to the infant sleep environment
  Interventions: Behavioral: Reduce Infant Mortality

INTERVENTIONS:
Behavioral: Reduce Infant Mortality — The study's long term goal is to disseminate a new easily implemented and reproducible intervention that based on our previous research is culturally competent and provides a rationale for changing infant sleep position and sleep environment. This intervention if successful will quickly be disseminated and will be an important change to the system of newborn care; the resultant change in parental behavior would ultimately result in a reduction in sleep-related infant mortality rates thereby promoting healthy development.After written consent has been obtained, a brief survey about knowledge of and attitudes toward safe sleep position recommendations, current intent with regards to safe sleep recommendations, and demographics will be completed. Contact information will be obtained from participants to facilitate study follow-up at two weeks of infants birth 2-3 months and 5-6 months.
  Other Names: African Americans; Anticipatory guidance; Health Promotion; Infant Mortality; Injury Prevention; Nurses; Parent Education; Sudden Infant Death Syndrome

SUMMARY:
The overall purpose of this randomized trial is to develop and evaluate a systematic approach to improve African-American parental behaviors specifically with regards to the infant sleep environment. African-American parents of newborn, healthy term infants will be randomized to receive either a standard message to avoid bedsharing, eliminate use of soft bedding and soft sleep surfaces, and to place infants in the supine position for sleep to reduce the risk of SIDS or an enhanced message to avoid these behaviors to both reduce the risk of SIDS and to prevent infant suffocation.

DETAILED DESCRIPTION:
A persistent, significant racial disparity exists in infant mortality rates attributable to Sudden Infant Death Syndrome (SIDS) and other types of sleep-related sudden unexpected infant death (SUID), such as suffocation and undetermined causes of death. SIDS and other sleep-related deaths account for ~4600 U.S. deaths annually.4 While the incidence of SIDS has declined, infant deaths from accidental suffocation and strangulation in bed have quadrupled.5 Additionally, racial disparities in SIDS and other sleep-related deaths have increased over the past decade, with African-American infants twice as likely to die as other infants.6, 7 Certain infant sleeping practices, such as prone (stomach) sleeping, use of soft bedding and soft sleep surfaces, and bedsharing, likely play a significant role, both in SIDS and SUID, and in the disparities seen therein. Elimination of health barriers and racial/ethnic disparities, and promoting healthy development, have been highlighted as MCHB research priorities; this application is directly responsive to both of these priorities.

In the current system, health care providers and public health messages, using the American Academy of Pediatrics (AAP) recommendations,8 stress the use of supine (back) positioning, avoidance of soft bedding, and room sharing without bedsharing as recommendations to reduce the risk of SIDS. However, our research suggests that African-Americans have problems with this message, as they have a low degree of self-efficacy with regards to SIDS risk reduction (i.e., they do not believe that their actions can make a difference in whether SIDS occurs) and are suspicious of the concept of "risk reduction."2 However, African-American parents have a high degree of self-efficacy with regards to preventing infant suffocation. Given the increasing number of suffocation and other preventable sleep-related deaths and the fact that many of the behavioral risk factors for both SIDS and preventable sleep-related deaths are the same, providing parents with an additional safe sleep message that emphasizes prevention of suffocation may be more effective in changing parent behavior. Such a message would be carefully crafted based on our current community-based research1-3 to address emerging risks of greatest concern and potential self-efficacy. A simple, easily reproducible change in the system of newborn care could thus address a critical barrier to further progress in reducing infant mortality rates, particularly among African American families. The best systems of care to reduce disparities must use the best available and culturally competent messaging based on strong empirical evidence and require rigorous evaluation.

ELIGIBILITY:
Inclusion Criteria:

* The purpose of the study is to determine the impact of a new educational strategy on African American parents, all participants will be self identified as African American. Although male parents will be allowed to participate in the followup surveys, female parents will be the primary focus of this study.

Exclusion Criteria:

* Mothers under the age of 18 years will not be included in the study. Infants born with congenital anomalies that would prevent them from sleeping in the supine position or if the infant is born at less than 36 weeks gestation, requires hospitalization for more than 1 week, or has ongoing medical problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2011-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Suffocation, Strangulation and Sudden Infant Death Syndrome | Three years
  Sleep Position (Supine vs. Nonsupine) Bedsharing (Yes vs. No) Use of Softbedding (Yes vs. No)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Y Moon, MD, Principal Investigator — University of Virginia
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Moon RY, Mathews A, Joyner BL, Oden RP, He J, McCarter R. Health Messaging and African-American Infant Sleep Location: A Randomized Controlled Trial. J Community Health. 2017 Feb;42(1):1-9. doi: 10.1007/s10900-016-0227-1. PMID 27470122
- [Derived] Mathews A, Joyner BL, Oden RP, He J, McCarter R Jr, Moon RY. Messaging Affects the Behavior of African American Parents with Regards to Soft Bedding in the Infant Sleep Environment: A Randomized Controlled Trial. J Pediatr. 2016 Aug;175:79-85.e2. doi: 10.1016/j.jpeds.2016.05.004. Epub 2016 Jun 2. PMID 27263400